CLINICAL TRIAL: NCT04173572
Title: Targeting Physical Health in Schizophrenia: Physical Activity Can Enhance Life Randomized Control Trial
Acronym: (PACE-life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-2286; 1R34MH111852-01A1 (NIH)
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Results first posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Brief Psychotic Disorder; Schizophreniform Disorders; Unspecified Schizophrenia Spectrum and Other Psychotic Disorder
Keywords: Walking; Exercise; Physical Health
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking Group (Experimental): Participants will be walking two times a week in supervised virtual walking groups on a secure online platform (Zoom) and will also participate in independent walks done at a location of their own choosing outside group participation.
  Interventions: Behavioral: PACE-Life
- Fitbit Alone (Active Comparator): Participants will be provided with a Fitbit wristband and instructed how to use it. Participants will also be given information on current recommended physical activity guidelines and told that study staff may be contacting them on a weekly basis if it looks like participants are not wearing their Fitbit for a certain number of days or to troubleshoot any issues.
  Interventions: Behavioral: Exercise Intervention

INTERVENTIONS:
Behavioral: PACE-Life — PACE-Life Groups will occur twice per week for 15 minutes in the first two weeks, progressing to 30-minute walking sessions over the course of the intervention without changes in frequency. The intensity of virtual walks will increase throughout this intervention in a stepwise fashion to create an exercise dose response to maximize impact on CRF.
  Other Names: Exercise Intervention
  Arms: Walking Group
Behavioral: Exercise Intervention — Data from Fitbit devices will be synced and accessed through Fitbit.com. Participants will be provided account information to view data but will be asked not to change any of the settings as the investigators will be using data for tracking steps/day and minutes spent walking.
  Other Names: Fitbit
  Arms: Fitbit Alone

SUMMARY:
Purpose: To test the effectiveness of an exercise intervention that combines group walking, activity tracking, and heart rate monitoring (i.e. Physical Activity can Enhance Life, PACE-Life) on the physical and mental health for individuals with schizophrenia spectrum disorder.

Participants: 50 individuals with schizophrenia spectrum disorders.

Procedures (methods): During the baseline assessment, which can be completed virtually and in-person (based on participant preference) all participants will be provided with a Fitbit wristband and instructed how to use it. During the first group session, participants will be taught how to use their heart rate (on the Fitbit) to determine how fast participants should walk (to achieve the appropriate exercise dosage). Information on proper care, usage, and how to determine the appropriate heart rate from the watch, to guide the intensity of the walk, will be provided to participants and reviewed at each group session. Participants randomly assigned to the PACE Life virtual walking group sessions will meet the other group members and group leaders and be reminded of the heart rate (HR) that corresponds with the intensity of that group session. Next, the group will exercise for 15 minutes in the first two weeks, progressing to 30-minute walking sessions over the course of the intervention. At the completion of the sessions, everyone will take a break for water and review the walk. After the second group session of each week, participants will receive weekly progress reports of their steps and minutes spent walking the prior week (obtained from Fitbit devices). During this session, participants will also set individual goals for the upcoming week for both their "intensity walks" and total steps per day.

Participants randomly assigned to Fitbit Alone will be given a Fitbit and shown how to use it by study staff. Participants will also be given information on current recommended physical activity guidelines (150 min/week of moderate intensity exercise) and will be told that study staff may be contacting them on a weekly basis (or shorter, if necessary) if it looks like participants are not wearing their Fitbit for a certain number of days (e.g. 3 consecutive days) or to troubleshoot any issues. If necessary, participants might be invited to meet with research staff to get assistance on any Fitibit or exercise-related issues.

DETAILED DESCRIPTION:
Overview of Procedures: The PACE-Life Group will be integrated into the Schizophrenia Treatment and Evaluation Program (STEP) outpatient clinics in Raleigh, NC and Carrboro, NC. The group walks will occur on a secure online platform (Zoom). Goal-setting groups and all assessments will also take place on a secure online platform (Zoom). Goal-setting will include setting goals for the upcoming week in terms of number of steps as well as how many intensity walks individuals plan to complete. Clinic-based group sessions will also include if-then plans and problem solving any issues that interfere with home-based walks.

The Fitbit Alone participants will be given a Fitbit and instructed on how to use them as well as information on current recommended physical activity guidelines. Participants will be told that study staff may be contacting them on a weekly basis (or shorter, if necessary) if it looks like they are not wearing their Fitbit for a certain number of days or to troubleshoot any issues. If necessary participants may be invited to meet with research staff to receive assistance on any Fitbit or exercise-related issues.

Assessments/Measures: The exercise intervention, PACE-Life, will last for 16 weeks and includes both virtual group walks and independent walks. Participants will be asked to complete assessments (either virtually or in-person based on preference) at screening, baseline, mid-point, post-test, and 1-month follow-up.

At Screening the following measures will be examined: Demographics, the Wide Range Achievement Test (WRAT), a licensed physician will complete a medical history and physical exam to provide medical clearance for participants, Physical Activity Readiness Questionnaire (PAR-Q) and the -the Mini-International Neuropsychiatric Interview (MINI) will be used to verify that participants have a schizophrenia spectrum diagnosis before they are enrolled in the study.

At the Baseline, Mid-point, Post-test, and 1-Month Follow-up the following measures will be examined: Demographics, Minutes Spent Walking, the Short Form International Physical Activity Questionnaire (IPAQ), Steps/day, Cardiorespiratory fitness (CRF)- CRF will be measured using the 6-minute walk test (6MWT), if in person, or compute CRF based on an equation by Jackson, A.S., et al (1990) that includes recent weight and height, for the calculation of BMI, gender, self-reported physical activity level, and age, Self-determination Basic Needs, the Basic Psychological Need Scale-in General, the Basic Psychological Needs in Exercise Scale (BPNES), the Positive and Negative Syndrome Scale (PANSS), Resting Systolic/Diastolic Blood Pressure and resting heart rate (RHR), autonomous motivation will be measured with the Behavioral Regulation in Exercise Questionnaire-2 (BREQ-2), enjoyment of walking will be measured with the Physical Activity Enjoyment Scale (PACES), the UCLA Loneliness Scale, Weight, BMI, and Waist/hip Circumference.

At the conclusion of the open trial, the investigators will administer a brief questionnaire to the participants regarding satisfaction and acceptability that will include both Likert ratings and open-ended questions.

Intervention- PACE-Life Groups will occur twice per week for 15 minutes in the first two weeks, progressing to 30-minute walking sessions over the course of the intervention without changes in frequency. The intensity of virtual walks will increase throughout the intervention in a stepwise fashion to create an exercise dose response to maximize impact on CRF.

Fitbits: All participants will be provided a Fitbit that is labeled with a participant number. All Fitbits are paired to a Fitbit account. Data from Fitbit devices can be synced to the corresponding account and accessed through Fitbit.com. Participants will be provided information about their accounts should participants want to look at the data but will be asked not to change any of the settings as the investigators will be using data for tracking steps/day and minutes spent walking.

Protocol Changes due to COVID-19 Pandemic:

Protocol changes due to the COVID-19 pandemic have been formalized and made permanent as outlined above. Additionally, walking groups will take place virtually, on a secure online platform (Zoom). The Wide Range Achievement Test (WRAT) will be used instead of the Wechsler Abbreviated Scale of Intelligence (WASI) to measure a minimum reading level (4th grade) to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* DSM-V diagnosis of a SSD (Schizophrenia, Schizoaffective Disorder, Brief Psychotic Disorder, Schizophreniform Disorder, and Unspecified Schizophrenia Spectrum and Other Psychotic Disorder)
* Between the ages of 18-65, both genders, and any ancestry
* Reading level > 4th grade. Reading level will be measured by WRAT.
* No hospitalizations for psychiatric reasons in the last 3 months
* Clinically stable (no psychiatric medication changes within the past month)
* Are not already engaging in consistent moderate-intensity exercise (cutoff = 60 min/week for the past 6 months)
* Present with no contra-indication to engage in regular moderate intensity exercise based on the American College of Sports Medicine guidelines
* Willing and able to provide informed consent or has legal guardian present to provide informed consent.

Exclusion Criteria:

* Pregnant women will be excluded because pregnancy alters autonomic and immune responsiveness, increase weight gain, and can influence heart rate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L Penn, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - North Carolina Psychiatric Research Center, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: 9 to 36 months following publication
Access Criteria: Requesting investigator has appropriate approval (see above) and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomly assigned to a group by an unblinded research assistant after they were screened as eligible and created a baseline appointment time with the research coordinator.
Period: Overall Study
Arm/Group | Walking Group | Fitbit Alone
Started | 24 | 26
Cohort 1 | 7 | 6
Cohort 2 | 8 | 12
Cohort 3 | 9 | 8
Completed | 20 | 20
Not Completed | 4 | 6
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Walking Group | Fitbit Alone | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Full Range); unit: years] | 40.38 [22 to 62] | 39.89 [21 to 62] | 40.14 [21 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 10 | 15 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 20 | 25 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 11 | 16 | 27
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 26 | 50
Occupation [Count of Participants; unit: Participants]
  Employed | 7 | 4 | 11
  Unemployed/Disability | 17 | 16 | 33
  Student | 0 | 6 | 6
MINI - Psychotic Disorders [Count of Participants; unit: Participants] — MINI International Neuropsychiatric Interview (MINI) is a brief structured diagnostic interview and is designed to assess the most common psychiatric disorders in ICD-10 and DSM-5. MINI modules were used: mood disorders with psychotic features, psychotic disorders. Questions are rated dichotomously (yes/no) and clinical judgment should be used in coding the responses, asking for examples if needed. Participants will be eligible for the study if they are diagnosed with a lifetime or current psychotic disorder based on the MINI assessment.
  Participants
    Lifetime mood disorder w/ psychotic features | 2 | 2 | 4
    Current mood disorder w/ psychotic features | 0 | 0 | 0
    Lifetime psychotic disorder | 22 | 25 | 47
    Current psychotic disorder | 13 | 13 | 26
WRAT 3 Word Reading Task (Raw Score) [Mean (Standard Deviation); unit: units on a scale] — The WRAT 3 Reading task measures intellectual ability level through word and letter recognition. This task provides participants with a list of progressively difficult words to read aloud to the tester. 42 words are provided to the participant on the sheet of paper from which they are asked to read. Each word read aloud correctly earns the participant 1 point. Scores range between 0 and 42, with higher scores indicating higher abilities and achievements. Participants were required to read 32 words correctly (equivalent to a fourth grade reading level) to be eligible for the study. Population: This data was not collected during cohort 1 of the trial.
  units on a scale
    number analyzed (Participants) | 17 | 20 | 37
    (all) | 36.24 (3.49) | 37.05 (3.09) | 36.65 (3.23)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Participant's Total Distance During 6-minute Walk
Description: The 6-minute walk test (6MWT) will be used to measure cardiorespiratory fitness (CRF) during which individuals will be asked to walk continuously for six minutes on a flat, indoor surface around cones (separated by 100ft). The possible distance range is 400 meters to 650 meters. Higher scores reflect better outcomes (greater physical fitness).
Time Frame: Baseline and the last study visit (Up to 20 weeks)
Population: Participants were only analyzed from cohorts 2 and 3 as cohort 1 was deemed not comparable (protocol changes & cancellation after 7 groups due to the onset of the COVID-19 pandemic). Participants who completed assessments from home were unable to provide data on this measure (n=5 in walking group, n=9 in fitbit alone). Post-treatment data are not available for participants who withdrew or were lost to follow-up (n=1 in walking group, n=2 in Fitbit alone).
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Walking Group | Fitbit Alone
Number analyzed (Participants) | 12 | 11
meters
  Baseline | 458.775 (91.467) | 467.209 (83.828)
  Post-treatment: number analyzed (Participants) | 11 | 9
  Post-treatment | 452.355 (103.346) | 448.711 (59.594)
Statistical Analysis 1: Comparison: Walking Group; Posttreatment - Baseline: 10 participants analyzed (had data at both time points); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = -13.470, Standard Deviation 48.09
Statistical Analysis 2: Comparison: Fitbit Alone; Posttreatment - Baseline: 9 participants analyzed (had data at both time points); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = 1.700, Standard Deviation 52.743

2. Secondary Outcome: Mean Difference in Minutes Spent Walking
Description: Mean difference in overall minutes spent walking per week from baseline to last study visit (up to 20 weeks). This information will be obtained from the participant's Fitbit. Higher scores reflect more minutes walking.
Time Frame: Baseline and the last study visit (up to 20 weeks)
Population: Participants were only analyzed from cohorts 2 and 3 as cohort 1 was deemed not comparable (protocol changes & cancellation after 7 groups due to the onset of the COVID-19 pandemic). Data was not available from all participants as it was dependent upon consistent daily wearing of Fitbit device. Post-treatment data are not available for participants who withdrew or were lost to follow-up (n=2 in walking group, n=2 in Fitbit alone).
Measure: Mean (Standard Deviation); unit: minutes/week
Arm/Group | Walking Group | Fitbit Alone
Number analyzed (Participants) | 17 | 18
minutes/week
  Baseline | 31.647 (40.812) | 44.278 (88.842)
  Post-treatment: number analyzed (Participants) | 15 | 16
  Post-treatment | 55.866 (83.874) | 58.188 (149.560)
Statistical Analysis 1: Comparison: Walking Group; Posttreatment - Baseline: 15 participants analyzed (had data at both time points); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = 22.133, Standard Deviation 79.938
Statistical Analysis 2: Comparison: Fitbit Alone; Posttreatment - Baseline: 15 participants analyzed (had data at both time points); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = 7.80, Standard Deviation 99.645

3. Secondary Outcome: Mean Difference in Daily Steps
Description: Mean difference in daily steps from baseline to last study visit (up to 20 weeks). This information will be obtained from the participants Fitbit. Higher scores reflect more daily steps.
Time Frame: Baseline and the last study visit (Up to 20 weeks)
Population: Participants were only analyzed from cohorts 2 and 3 as cohort 1 was deemed not comparable (protocol changes & cancellation after 7 groups due to the onset of the COVID-19 pandemic). Data was not available from all participants as it was dependent upon consistent daily wearing of Fitbit device. Post-treatment data are not available for participants who withdrew or were lost to follow-up (n=3 in walking group, n=2 in Fitbit alone).
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | Walking Group | Fitbit Alone
Number analyzed (Participants) | 17 | 18
steps/day
  Baseline | 4940.529 (4463.869) | 5010.667 (3487.757)
  Post-treatment: number analyzed (Participants) | 14 | 16
  Post-treatment | 4274.429 (3039.565) | 4503.875 (3860.307)
Statistical Analysis 1: Comparison: Walking Group; Posttreatment - Baseline: 14 participants analyzed (had data at both time points); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = 13.642, Standard Deviation 4213.837
Statistical Analysis 2: Comparison: Fitbit Alone; Posttreatment - Baseline: 15 participants analyzed (had data at both time points); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = -483.4, Standard Deviation 2497.312

4. Secondary Outcome: Mean Difference Overall UCLA Loneliness Scale Score
Description: Mean difference in overall score from baseline to last study visit (up to 20 weeks). The UCLA Loneliness scale is a 20 item scale. Answers are on a 4 point scale with options "I often feel this way," "I sometimes feel this way," "I rarely feel this way," and "I never feel this way." Possible scores range from 20 to 80. Higher scores reflect worse outcomes (greater feelings of loneliness).
Time Frame: Baseline and the last study visit (Up to 20 weeks)
Population: Participants were only analyzed from cohorts 2 and 3 as cohort 1 was deemed not comparable (protocol changes & cancellation after 7 groups due to the onset of the COVID-19 pandemic). Post-treatment data are not available for participants who withdrew or were lost to follow-up (n=2 in walking group, n=4 in Fitbit alone).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Walking Group | Fitbit Alone
Number analyzed (Participants) | 17 | 20
score on a scale
  Baseline | 48.588 (11.979) | 46.450 (11.353)
  Post-treatment: number analyzed (Participants) | 15 | 16
  Post-treatment | 50.133 (10.370) | 47.812 (11.485)
Statistical Analysis 1: Comparison: Walking Group; Posttreatment - Baseline: 15 participants analyzed (had data at both time points); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = -0.800, Standard Deviation 4.229
Statistical Analysis 2: Comparison: Fitbit Alone; Posttreatment - Baseline: 16 participants analyzed (had data at both time points); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = 1.563, Standard Deviation 8.695

5. Secondary Outcome: Mean Difference Overall PANSS Score
Description: Mean difference in the overall score from baseline to last study visit (up to 20 weeks). The PANSS is a semi-structured interview using a 30-item scale to evaluate the presence, absence and severity of Positive, Negative and General Psychopathology symptoms of schizophrenia. All 30 items are rated on a 7-point scale (1 = absent; 7 = extreme). Possible scores range from 30 to 210. Higher scores reflect worse outcomes (i.e. greater symptoms of psychosis).
Time Frame: Baseline and the last study visit (Up to 20 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Walking Group | Fitbit Alone
Number analyzed (Participants) | 17 | 20
score on a scale
  Baseline | 62.588 (12.227) | 60.700 (9.183)
  Post-treatment: number analyzed (Participants) | 15 | 16
  Post-treatment | 55.467 (9.211) | 61.062 (14.289)
Statistical Analysis 1: Comparison: Walking Group; Posttreatment - Baseline: 15 participants analyzed (had data at both time points); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Median Difference (Net) = -9.333, Standard Deviation 14.166
Statistical Analysis 2: Comparison: Fitbit Alone; Posttreatment - Baseline: 16 participants analyzed (had data at both time points); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Median Difference (Net) = 0.625, Standard Deviation 9.664

6. Secondary Outcome: Mean Difference in Body Mass Index (BMI) Change
Description: Mean difference in BMI from baseline to last study visit (up to 20 weeks). Expected normal BMI ranges from 14 to 54. Higher scores reflect worse outcomes (i.e., greater body mass).
Time Frame: Baseline and the last study visit (Up to 20 weeks)
Population: Participants were only analyzed from cohorts 2 and 3 as cohort 1 was deemed not comparable (protocol changes & cancellation after 7 groups due to the onset of the COVID-19 pandemic). Some participants who completed assessments from home were unable to provide accurate data on this measure (n=2 in walking group, n=2 in fitbit alone). Post-treatment data are not available for participants who withdrew or were lost to follow-up (n=2 in Fitbit alone).
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Walking Group | Fitbit Alone
Number analyzed (Participants) | 15 | 18
kg/m^2
  Baseline | 36.026 (8.296) | 36.872 (9.819)
  Post-treatment: number analyzed (Participants) | 15 | 16
  Post-treatment | 33.553 (6.764) | 36.262 (11.183)
Statistical Analysis 1: Comparison: Walking Group; Posttreatment - Baseline: 13 participants analyzed (had data at both time points); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = -0.392, Standard Deviation 1.148
Statistical Analysis 2: Comparison: Fitbit Alone; Posttreatment - Baseline: 15 participants analyzed (had data at both time points); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = .113, Standard Deviation 1.401

7. Secondary Outcome: Mean Difference in Body Weight Change
Description: Mean difference in body weight change from baseline to last study visit (up to 20 weeks).
Time Frame: Baseline and the last study visit (Up to 20 weeks)
Population: Participants were only analyzed from cohorts 2 and 3 as cohort 1 was deemed not comparable (protocol changes & cancellation after 7 groups due to the onset of the COVID-19 pandemic). Some participants who completed assessments from home were unable to provide accurate data on this measure (n=2 in fitbit alone). Post-treatment data are not available for participants who withdrew or were lost to follow-up (n=2 in walking group, n=3 in Fitbit alone).
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Walking Group | Fitbit Alone
Number analyzed (Participants) | 17 | 18
lbs
  Baseline | 228.11 (60.56) | 240.88 (66.43)
  Post-treatment: number analyzed (Participants) | 15 | 15
  Post-treatment | 220.96 (47.62) | 235.75 (74.29)
Statistical Analysis 1: Comparison: Walking Group; Posttreatment - Baseline: 15 participants analyzed (had data at both time points); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = 2.20, Standard Deviation 20.11
Statistical Analysis 2: Comparison: Fitbit Alone; Posttreatment - Baseline: 15 participants analyzed (had data at both time points); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = 0.49, Standard Deviation 8.91

8. Secondary Outcome: Mean Difference in Waist Circumference
Description: Mean difference in waist circumference from baseline to last study visit (up to 20 weeks). Higher scores reflect worse outcomes.
Time Frame: Baseline and the last study visit (Up to 20 weeks)
Population: Participants were only analyzed from cohorts 2 and 3 as cohort 1 was deemed not comparable (protocol changes & cancellation after 7 groups due to the onset of the COVID-19 pandemic). Some participants who completed assessments from home were unable to provide accurate data on this measure (n=4 in walking group, n=7 in fitbit alone). Post-treatment data are not available for participants who withdrew or were lost to follow-up (n=1 in walking group, n=2 in Fitbit alone).
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Walking Group | Fitbit Alone
Number analyzed (Participants) | 13 | 13
cm
  Baseline | 109.88 (18.58) | 112.30 (20.82)
  Post-treatment: number analyzed (Participants) | 12 | 11
  Post-treatment | 106.94 (17.54) | 115.94 (27.36)
Statistical Analysis 1: Comparison: Walking Group; Posttreatment - Baseline: 11 participants analyzed (had data at both time points); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = -0.39, Standard Deviation 4.67
Statistical Analysis 2: Comparison: Fitbit Alone; Posttreatment - Baseline: 11 participants analyzed (had data at both time points); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = 3.43, Standard Deviation 9.4

9. Secondary Outcome: Mean Difference in Systolic Blood Pressure Change
Description: Mean difference in systolic blood pressure change from baseline to last study visit (up to 20 weeks).
Time Frame: Baseline and the last study visit (Up to 20 weeks)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Walking Group | Fitbit Alone
Number analyzed (Participants) | 17 | 18
mmHg
  Baseline | 125 (9.663) | 129.167 (8.333)
  Post-treatment: number analyzed (Participants) | 15 | 15
  Post-treatment | 122 (9.878) | 124.867 (12.047)
Statistical Analysis 1: Comparison: Walking Group; Posttreatment - Baseline: 15 participants analyzed (had data at both time points); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = -3.667, Standard Deviation 9.067
Statistical Analysis 2: Comparison: Fitbit Alone; Posttreatment - Baseline: 14 participants analyzed (had data at both time points); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = -2.071, Standard Deviation 12.250

10. Secondary Outcome: Mean Difference in Diastolic Blood Pressure Change
Description: Mean difference in diastolic blood pressure change from baseline to last study visit (up to 20 weeks).
Time Frame: Baseline and the last study visit (Up to 20 weeks)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Walking Group | Fitbit Alone
Number analyzed (Participants) | 17 | 18
mmHg
  Baseline | 77.647 (8.746) | 81.111 (10.459)
  Post-treatment: number analyzed (Participants) | 15 | 15
  Post-treatment | 76.000 (9.921) | 78.533 (13.174)
Statistical Analysis 1: Comparison: Walking Group; Posttreatment - Baseline: 14 participants analyzed (had data at both time points); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = -0.800, Standard Deviation 9.900
Statistical Analysis 2: Comparison: Fitbit Alone; Posttreatment - Baseline: 14 participants analyzed (had data at both time points); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = 0.714, Standard Deviation 11.717

11. Secondary Outcome: Mean Difference in Resting Heart Rate Change
Description: Mean difference in resting heart rate change from baseline to last study visit (up to 20 weeks). Expected normal heart rate ranges from 40 to 120. Higher scores reflect worse outcomes (poorer heart condition).
Time Frame: Baseline and the last study visit (Up to 20 weeks)
Population: Participants were only analyzed from cohorts 2 and 3 as cohort 1 was deemed not comparable (protocol changes & cancellation after 7 groups due to the onset of the COVID-19 pandemic). Some participants who completed assessments from home were unable to provide accurate data on this measure (n=1 in walking group, n=4 in fitbit alone). Post-treatment data are not available for participants who withdrew or were lost to follow-up (n=1 in walking group).
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Walking Group | Fitbit Alone
Number analyzed (Participants) | 16 | 16
beats per minute
  Baseline | 77.188 (12.319) | 77.313 (13.459)
  Post-treatment: number analyzed (Participants) | 15 | 16
  Post-treatment | 82.133 (10.548) | 80.625 (8.966)
Statistical Analysis 1: Comparison: Walking Group; Posttreatment - Baseline: 14 participants analyzed (had data at both time points); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = 3.071, Standard Deviation 10.737
Statistical Analysis 2: Comparison: Fitbit Alone; Posttreatment - Baseline: 14 participants analyzed (had data at both time points); Test type: Other — Single group mean difference between baseline and post-treatment assessments; Mean Difference (Net) = 5.571, Standard Deviation 9.288

12. Other Pre Specified Outcome: Mean Difference in Composite Motivation Score on the Behavioral Regulation Exercise Questionnaire (BREQ-2)
Description: Mean difference in composite motivation score from baseline to last study visit (up to 20 weeks). The BREQ-2 is a 19 item self-report scale. Answers are on a 5 point Likert scale ranging from 0 to 4. 0 corresponds to "not true for me" and 4 corresponds to "very true for me." Possible scores are averaged and range from 0-4. Higher scores reflect better outcomes (higher autonomous motivation to exercise).
Time Frame: Baseline and the last study visit (Up to 20 weeks)
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Mean Difference in Composite Score on the Basic Psychological Needs in Exercise Scale (BPNES)
Description: Mean difference in composite score from baseline to last study visit (up to 20 weeks). The BPNE is an 11 item self-report scale. Answers are on a 5 point Likert scale ranging from "I don't agree at all" to "I completely agree." Possible scores are averaged and range from 1-5. Higher scores reflect better outcomes (i.e. more psychological needs being met through exercise).
Time Frame: Baseline and the last study visit (Up to 20 weeks)
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Mean Difference in Composite Score on the Physical Activity Enjoyment Scale (PACES)
Description: Mean difference in composite score from baseline to last study visit (up to 20 weeks). 2. The PACES is an 18 item self-report scale. Answers are on a 7-point scale. Possible scores are averaged and range from 1-7. Higher scores reflect better outcomes (greater enjoyment of physical activity).
Time Frame: Baseline and the last study visit (Up to 20 weeks)
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Mean Difference in Composite Score on the Basic Psychological Needs Scale (BPNS)
Description: Mean difference in composite score from baseline to last study visit (up to 20 weeks). The BPNS is a 21 item self-report scale. Answer are on a 7-point Likert scale ranging from "not at all true" to "very true." Possible scores on each subscale are averaged onto a scale of 1-7. Higher scores reflect better outcomes (better autonomy, competence, and relatedness).
Time Frame: Baseline and the last study visit (Up to 20 weeks)
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Mean Difference in Composite Score on the Autonomy Support Scale
Description: Mean difference in composite score from mid-treatment to last study visit (up to 20 weeks). The Autonomy Scale is a 6 item self-report scale. Answers are made using a 7-point scale. Possible scores range from 7 to 46. Higher scores reflect better outcomes (better relationship between research participant and staff.
Time Frame: Baseline and the last study visit (Up to 20 weeks)
Reporting Status: Not Posted

17. Other Pre Specified Outcome: End of Study Survey
Description: Total score at Post treatment visit only (16 weeks). The End of Study survey measures participant's satisfaction and feedback with the PACE-Life trial. The survey is a 18 item self-report scale, consisting of both Likert scale and open-ended items. Answers are made using a 5-point Likert scale. Possible scores on each item range from 1-5. Higher scores reflect higher levels of satisfaction and enjoyment in the study.
Time Frame: Post treatment only (16 weeks)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent by each subject until they completed study procedures, for a duration of up to 20 weeks for each subject.
Arm/Group | Walking Group | Fitbit Alone
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/24 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Walking Group (N=24) | Fitbit Alone (N=26)
Hospitalization unrelated to study (Psychiatric disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This trial began in early 2020, immediately before the onset of the COVID-19 pandemic. As such, the 13 participants in cohort 1 did not have complete trial data. Cohorts 2 and 3 were later run virtually. While a total of 50 participants were enrolled, only 37 of those participants were analyzed as the first 13 participants created data that was deemed unusable and incomparable to the data from cohorts 2 and 3.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/72/NCT04173572/Prot_SAP_000.pdf